CLINICAL TRIAL: NCT06568601
Title: Reducing Veterans' Risk of Atherosclerotic Cardiovascular Disease Through Pharmacogenomics Informed Statin Prescribing
Brief Title: Pharmacogenomic Informed Statin Prescribing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 21-040; I01HX003477-01A3 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hypercholesterolemia
Keywords: Atherosclerosis; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Pharmacogenomic Testing; Genetic Risk Score
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis; Genetic Risk Score | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Patient randomized, open-label, parallel group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Genetic testing arm (Experimental): The intervention involves: genetic testing; interpretation; and prior to and shortly following an upcoming appointment, communication to patients and providers about the patients' predicted statin efficacy and toxicity, genetic risk for CVD, and individualized recommended statin type/dose.
  Interventions: Genetic: Pharmacogenetic and polygenic risk testing
- Control (Active Comparator): The control condition involves receipt of a report highlighting the risk of cardiovascular disease and benefits of statins (without genetic test results).
  Interventions: Other: Active control

INTERVENTIONS:
Genetic: Pharmacogenetic and polygenic risk testing — The intervention involves: genetic testing; interpretation; and prior to and shortly following an upcoming appointment, communication to patients and providers about the patients' predicted statin efficacy and toxicity, genetic risk for CVD, and individualized recommended statin type/dose.
  Arms: Genetic testing arm
Other: Active control — The control condition involves receipt of a report highlighting the risk of cardiovascular disease and benefits of statins (without genetic test
  Other Names: Control
  Arms: Control

SUMMARY:
Statins are the most cost-effective medications to lower cholesterol and cardiovascular disease (CVD) risk. However, many patients at high-risk for CVD do not accept or adhere to statins. This gap in patient's use of statins limits the full impact of these effective medications resulting in higher cholesterol levels and CVD risk. The main barriers to using statins are patients' perceived lack of benefit, excess risk of statin toxicity as well as their misperceptions of their CVD risk. Statin pharmacogenomic testing - an application of precision medicine - is a readily available, feasible, and inexpensive intervention that addresses this barrier by using genetic testing to identify the nearly 1 out of 2 patients with enhanced benefit and/or reduced risk of statin toxicity or increased risk for CVD. By communicating statin pharmacogenomic test results to Veterans at high-risk for CVD not taking statin therapy, the investigators aim to improve patients' perceptions of their risk of CVD and statins and, in turn, their acceptance of and adherence to statins to reduce their cholesterol levels and CVD risk.

DETAILED DESCRIPTION:
Background: Despite the proven efficacy and safety of statins, nearly 250,000 Veterans at high-risk for cardiovascular disease (CVD) seen annually in primary care are not taking them leading to higher cholesterol levels, cardiovascular risk, and health care costs. Primary care providers and health systems have a critical and unmet need for pragmatic, scalable interventions to address gaps in their patients' perceptions of the risks and benefits of statin therapy to improve appropriate statin utilization and to lower CVD risk. Important prior work by the investigators group demonstrates that pharmacogenomic testing for statin toxicity is feasible, improves patients' perceptions of statin therapy, leads to a doubling in appropriate statin prescribing, and lowers cholesterol levels. The central hypothesis of this proposal is that disclosure of statin pharmacogenomic test results for statin efficacy/toxicity and CVD risk to patients at high-risk for CVD will improve their perceptions of their CVD risk and statins risks/benefits and, in turn, the proportion of Veterans accepting and adhering to statin therapy to achieve a clinically significant low-density lipoprotein cholesterol (LDL) reduction.

Significance: By using a feasible and inexpensive approach of pharmacogenomic testing for common genetic variants reporting on statin efficacy and toxicity and CVD risk, the work is significant as it will lead to more patients at high-risk for CVD accepting and adhering to statins. This work addresses HSR&D research priorities of quality and safety of health care and health care value, ORD priorities of increasing substantial real-world impact of VA research, and VHA quality measures around statin prescribing and controlling cholesterol levels in patients at high-risk for CVD.

Innovation and Impact: This proposal uses an innovative approach of pharmacogenomic testing to address patients' perceptions of the risks and benefits of statin therapy and their risk of CVD which are known barriers to statin acceptance and adherence. The investigators expect a positive impact on reducing CVD risk in Veterans.

Specific Aims:

1. Reduce cholesterol levels through a precision medicine approach of statin pharmacogenomic testing.
2. Improve acceptance of guideline-directed statin therapy through delivery of statin pharmacogenomic test results that communicates statin efficacy and toxicity.
3. Identify contextual and economic factors salient for implementing statin pharmacogenomic testing.

Methodology: A randomized controlled trial focused on effectiveness while secondarily gathering implementation data will enroll 408 primary care patients who are at high-risk for CVD and recommended for statins based on guidelines but not prescribed them. Participants will be randomized 1:1 to intervention (guideline-based statin recommendations - "guidelines" - plus statin pharmacogenomic test results) vs. control (guidelines) stratified by prior statin use. The primary outcome is change in 12-month LDL. Secondary outcomes are new statin prescriptions and patients' perceptions of risks and benefits of statins. Exploratory analyses will assess statin prescriptions and fills as potential mediators of the intervention. Qualitative data from trial participants and their providers will illuminate key factors to consider for future implementation. If effective, the cost-effectiveness and budget impact of the intervention on LDL during the trial period projected over 10-year and lifetime CVD risk horizons will be measured.

Next steps/Implementation: An embedded primary care, patient-powered caucus and a VA operational stakeholder board representing primary care, cardiology, pharmacy, and the VA Pharmacogenomics Testing for Veterans (PHASER) clinical program will work with the investigative team to create an implementation "blueprint" package consisting of patient/provider educational portfolios, electronic medical record tools, Corporate Data Warehouse queries, and laboratory protocols for dissemination to Veterans and VHA facilities.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the analysis if they:

* Are a Veteran
* Aged 40-75 years
* Diabetes mellitus or cardiovascular disease (coronary, cerebral, or peripheral artery disease)
* An upcoming primary care appointment in the next 4 months
* No active statin prescription (any time/dose, VA, or non-VA) in the prior 6 months
* English speaking
* At least 1 current active VA prescription
* At least 1 primary care appointment within the prior 2 years

Exclusion Criteria:

* Non-Veterans
* End-stage renal disease
* History of rhabdomyolysis
* Active treatment for non-dermatologic cancer
* Known, prior SLCO1B1 genetic test results
* Liver cirrhosis
* Palliative care or hospice in 1-year prior to admission, during hospital stay, or at discharge
* Active prescription for PCSK9 inhibitor
* Inability to provide informed consent due to language impairment, cognitive disease, or other similar factors at the discretion of the research assistant or project coordinator.
* Active enrollment in a different, interventional clinical trial, at the discretion of PI.
* History of allogeneic stem cell transplant or liver transplant.
* Documentation of specific adverse drug reactions thought to be attributed to statins:

  * Myopathy with associated elevation in creatinine kinase > 10x upper limit of normal
  * Angioedema
  * Elevated AST/ALT
  * Others at discretion of PI

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-07-28 (Estimated)

PRIMARY OUTCOMES:
Change in low density lipoprotein cholesterol | 15-months
  The primary effectiveness outcome will be the change in LDL-cholesterol level from baseline to 15-months.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Voora, MD, Principal Investigator — Durham VA Medical Center, Durham, NC; Dawn M. Bravata, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No